Effect of Monazite Sands in Patients with Osteoarthritis of the knee

Ethical committee Protocol No: 3.160.891

Telephone\_Contact\_Log

Documente date: May 3rd, 2019

## TELEPHONE CONTACT LOG

Effects of Sand Treatment on Osteoarthritis

| Official Title: Effect of Monazite Sands in Patients with Osteoarthritis of the Knee Ethical committee Protocol No: 3.160.891 Unique Protocol ID: T015-M02-2019AF00 | | | | | | F002 |
|---|---|---|---|---|---|---|
| S.No. | Date (dd/mm/yyyy) | Made call to | Purpose of the Call | Duration of the Call | Outcome of the<br>Matter Discussed | Signature of the personnel |
| Signature of the Principal Investigator: | | | | Date: | | |

**Study brief Title:**